CLINICAL TRIAL: NCT01462825
Title: The Protective Effect of Tomato Ketchup Consumption on Inflammation Induced Ex-vivo in Human Blood
Brief Title: The Effect of Tomato Ketchup on Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Antje Weseler, Principal Investigator, Maastricht University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: METC11-3-049
Record Dates: First submitted 2011-09-06; First posted 2011-10-31 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Inflammation
Keywords: Inflammation; cytokines; chemotaxis; tomatoes; cardiovascular disease
MeSH Terms: conditions — Inflammation; Chemotaxis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tomato ketchup meal (Experimental)
  Interventions: Dietary Supplement: tomato ketchup meal
- Placebo meal (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo meal

INTERVENTIONS:
Dietary Supplement: tomato ketchup meal — A single intake of 200 g tomato ketchup together with 200 g white cooked rice.
  Arms: tomato ketchup meal
Dietary Supplement: Placebo meal — Self-prepared vinaigrette matching the qualitative and quantitative macronutrient composition of the tomato ketchup together with 200 g cooked rice resulting in a meal that is isocaloric to the tomato-ketchup meal
  Arms: Placebo meal

SUMMARY:
The purpose of this study is to determine the inhibiting effects of a single consumption of tomato ketchup on inflammation which will be induced ex-vivo in human blood.

DETAILED DESCRIPTION:
The consumption of tomatoes and tomato products has been associated with a lower risk of developing cardiovascular disease and some types of cancer. Tomatoes and tomato products provide a good source of antioxidants (lipophilic and hydrophilic). The major tomato antioxidants comprise lycopene, α-tocopherol and ascorbic acid. It has been reported that these antioxidants in isolated form exert directly or indirectly anti-inflammatory effects in vitro. Studies with tomatoes or tomato products revealed that the observed anti-inflammatory effects could not be caused by the presence of only one antioxidant. It was suggested that these effects were due to the combination of antioxidants.

In recent cell culture studies with human endothelial cells we have shown that tomato ketchup exerts significant anti-inflammatory effects, which could be related to the particular composition of antioxidants, i.e. lycopene, ascorbic acid and α-tocopherol. Since, however, the relevance of the observed anti-inflammatory effects for humans is entirely unknown, the present pilot study aims to assess the acute effects of a single tomato ketchup consumption on ex vivo elicited inflammation in a small group of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 30 kg/m2
* Age >18 years

Exclusion Criteria:

* Occurence of any adverse event, in particular those which require the use of medication that might interfere with the effects and/or the uptake of the investigational products
* Intolerance of study products
* Occurence of a serious adverse event
* Use of supplements, functional foods and/or other products containing tomatoes, vitamins, antioxidants and polyphenolic compounds
* Use of a medically prescribed diet or slimming diet
* Vegetarian or vegan lifestyle
* Excessive alcohol consumption (< 28 consumptions (approximately 250 g alcohol) per week)
* Participation in a clinical trial within 4 weeks before the study
* Non-compliance with the demands of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Release of pro-and anti-inflammatory cytokines ex vivo | 2 months
  6h after consumption of tomato ketchup blood will be collected and challenged ex vivo with bacterial endotoxin (LPS) in order to elicit the release of pro- (TNF-alpha, IL-8) and anti-inflammatory cytokines (IL-10)

SECONDARY OUTCOMES:
Chemotaxis of monocytes ex vivo | 2 months
Antioxidant plasma concentrations | 2 months
  Quantification of lycopene, its stereoisomers, alpha-tocopherol, ascorbic acid in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Aalt Bast, Prof, PhD, Study Director — Maastricht University
Locations (1):
- Dept. of Toxicology, Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Background] Palozza P, Parrone N, Simone RE, Catalano A. Lycopene in atherosclerosis prevention: an integrated scheme of the potential mechanisms of action from cell culture studies. Arch Biochem Biophys. 2010 Dec 1;504(1):26-33. doi: 10.1016/j.abb.2010.06.031. Epub 2010 Jul 3. PMID 20599665
- [Background] Mateo Anson N, Aura AM, Selinheimo E, Mattila I, Poutanen K, van den Berg R, Havenaar R, Bast A, Haenen GR. Bioprocessing of wheat bran in whole wheat bread increases the bioavailability of phenolic acids in men and exerts antiinflammatory effects ex vivo. J Nutr. 2011 Jan;141(1):137-43. doi: 10.3945/jn.110.127720. Epub 2010 Nov 24. PMID 21106920
- [Background] Swennen EL, Bast A, Dagnelie PC. Immunoregulatory effects of adenosine 5'-triphosphate on cytokine release from stimulated whole blood. Eur J Immunol. 2005 Mar;35(3):852-8. doi: 10.1002/eji.200425423. PMID 15719372